CLINICAL TRIAL: NCT05501392
Title: South Texas Early Prevention Studies - PreK
Brief Title: South Texas Early Prevention Studies PreK
Acronym: STEPSPreK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Rio Grande Valley (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: STEPS
Record Dates: First submitted 2022-08-08; First posted 2022-08-15 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Childhood Obesity
Keywords: Prek children; obesity prevalence
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: There were three sequential data collection periods through the process.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors were blinded to study design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): This group received health education, P.E. classes, child nutritional services, as well as a parent component.
  Interventions: Behavioral: STEPS-PreK
- Control (Active Comparator): This group received their usual health education and P.E. classes.
  Interventions: Behavioral: STEPS-PreK

INTERVENTIONS:
Behavioral: STEPS-PreK — Intervention group received the BN CHSP, a Texas Education Agency (TEA)-approved CSHP. This health program was first piloted in schools located in low-income neighborhoods where enrollment was predominantly Black and Latino children. The Social-Ecological Model guided the BN CSHP design. This theory postulates that health behaviors are molded by individual, interpersonal, and environmental interactions. Thus, BN CSHP encompasses curricula from preschool to eighth grade and is designed to target the four environments that influence children's health behaviors: 1) Healthy Lifestyles Healthy Minds (Health), 2) Moving For Life (Physical Education), 3) Eat to Live (Child Nutrition/School Food Service), and 4) MyFamily/MiFamilia (Home).

SUMMARY:
The South Texas Early Prevention Study-Prekindergarten (STEPS-PreK4) was a cluster randomized trial (CRT) of preschool children 4 years of age to test the effect of the Bienestar/NEEMA Coordinated School Health Program (BN CSHP) on childhood obesity prevalence prevention.

DETAILED DESCRIPTION:
The STEPS-PreK4 was a CRT where preschools, embedded within elementary schools, were the unit of randomization, intervention, and analysis. The study was designed for two years of intervention (pre-kinder to kindergarten) and four data collection periods (fall 2018, spring 2019, fall 2019, and spring 2020). Due to the COVID-19 pandemic the study was stopped prematurely and only results from the first three periods will be presented.

The two school districts where the study was conducted are located along the Texas-Mexico border in the county of Hidalgo. These school districts were selected because of the high poverty and health risk-factors levels.25 The preschools have two grade levels with children 3 and 4 years of age. The present study targeted preschools with children 4 years of age. Demographics of the two school districts were similar, 99% Hispanic, 92% economically disadvantaged, and 42% identified as English as a second language.

ELIGIBILITY:
Inclusion Criteria:

* PreK children
* Enrolled in PSJA and La Joya ISDs

Exclusion Criteria:

* na

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1277 (Actual)
Dates: Start 2018-09-28 (Actual); Primary Completion 2020-03-17 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
cardiorespiratory fitness | 1.5 years
  as measured by the number of laps run in the Progressive Anaerobic Capacity Endurance Run (PACER) fitness test

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Alanis, Masters, Study Director — University of Texas Rio Grande Valley
Locations (1):
- University of Texas Rio Grande Valley, Edinburg, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Only aggregated data will be shared

REFERENCES:
- [Background] Trevino-Pena R, Wang X, Wang L, Romero Z, Alanis E, Li H. Social and Health Risk Factor Levels of Preschool Children Living Along the Texas-Mexico Border. J Sch Health. 2020 Dec 2. doi: 10.1111/josh.12979. Online ahead of print. PMID 33289119
- [Derived] Trevino-Pena R, Romero Z, Fuentes JC, Cortez KE, Alanis E, Alvarenga JCL. A Coordinated School Health Program Effect on Cardiorespiratory Fitness of South Texas Preschool Children: A Cluster Randomized Trial. J Sch Health. 2024 Apr;94(4):336-345. doi: 10.1111/josh.13414. Epub 2024 Jan 22. PMID 38252805
- See also: Website for STEPS PreK project protocol especially parental outreach newsletters and consent forms (English and Spanish). — https://www.utrgv.edu/stepsprek/

DOCUMENTS (3):
  • Study Protocol (2018-09-28): https://cdn.clinicaltrials.gov/large-docs/92/NCT05501392/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-28): https://cdn.clinicaltrials.gov/large-docs/92/NCT05501392/SAP_001.pdf
  • Informed Consent Form (2018-09-28): https://cdn.clinicaltrials.gov/large-docs/92/NCT05501392/ICF_002.pdf